CLINICAL TRIAL: NCT02779504
Title: Post Market Clinical Follow Up for the Evaluation of Reducing the Risk of Infection Using the Agluna® Treated METS Modular System
Brief Title: Post Market Clinical Follow Up Study for Evaluation of Agluna® METS
Status: Completed | Type: Observational
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-01
Record Dates: First submitted 2016-05-12; First posted 2016-05-20 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Agluna treated METS: Patient implanted with Agluna treated METS
- Untreated METS: Patient implanted with untreated METS

SUMMARY:
The Agluna® (antimicrobial ionic silver surface technology) is used to treat the surface of the METS (Modular Endoprosthetic Tumour System) medical devices, in order to reduce the risk of post surgical infections after orthopaedic endoprosthetic replacement surgery.

This Post Market Clinical Follow up study is designed to retrospectively establish the infection rate of a cohort patients who have received an Agluna® Treated METS implant and compare the clinical data to patients that have received an untreated METS implant; in order to provide evidence to support the investigators' clinical claims.

DETAILED DESCRIPTION:
This post-market clinical follow-up study will be a retrospective data comparison study of a series of Agluna® treated and untreated METS™ modular prostheses conducted at the Royal National Orthopaedic Hospital, Stanmore. The expected sample size will be 106, with 53 patients in each treatment arm (Agluna® treated vs untreated). However there will be an initial pilot of 20 subjects to evaluate the feasibility of the study conduct and to identify if any further study design modification are required.

The primary outcome is the estimation of the infection rate over 12 months following an Agluna (silver) treated METS™ endoprosthetic surgery. This will be compared to the infection rate of non-Agluna Treated devices in a similar population. Incidence of infection will be measured according to the accepted definition of periprosthetic joint infection from the American Academy of Orthopedic Surgeons. The study follow up period is 12 months after implantation. Secondary objectives are to examine the health economic impacts of using the Agluna® Treated METS™ Modular Tumour System in comparison to the untreated METS™ Modular Tumour System and to establish clinically relevant superiority of the Agluna® Treated METS™ Modular Tumour System in comparison to untreated METS™ Modular Tumour System.

ELIGIBILITY:
Inclusion Criteria:

1. Implanted with a METS™ modular implant at the Royal National Orthopaedic Hospital, Stanmore.
2. Patient was between 18 years old and 70 years old at the time of implantation.
3. Patient has been followed up for at least 12 months following implant surgery

Exclusion Criteria:

1. Patient is obese
2. Patient is currently or has been involved in pending litigation or worker's compensation
3. Patient has participated in another clinical investigation or study with an investigational medical device within the last 60 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female subjects aged between 18 years and 70 years who have been implanted with a METS™ modular implant at the Royal National Orthopaedic Hospital, Stanmore and the patient has been followed up for at least 12 months following implantation
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Infection rate in Agluna Treated METS in comparison to infection rate in untreated METs | Within 12 months following implantation of the METs implant
  The estimation of peri-prosthetic infection rate over twelve months following implantation with the Agluna® Treated METS™ Modular Tumour System. This will be compared to the infection rate of non- Agluna® Treated endoprostheses in a similar population.

SECONDARY OUTCOMES:
Health Economic Impacts of Agluna Treated METS versus Untreated METS will be examined by performing a cost analysis of the procedures | 12 months follow up post implantation
  To examine the health economic impacts of using the Agluna® Treated METS™ Modular Tumour System in comparison to the untreated METS™ Modular Tumour System, health economic questions will be addressed by analysing the costs of both treatments arms based on different models with varying assumptions for costs.
Superiority of the Agluna® Treated METS™ over the untreated METS for infection reduction will be established if the confidence interval lies below 0. | 12 months follow up post implantation
  To establish clinically relevant superiority of the Agluna® Treated METS™ Modular Tumour System in comparison to untreated METS™ Modular Tumour System, Investigation of superiority will be done analogously to the primary analysis. If the confidence interval lies completely below 0 superiority can be concluded. Additionally, to evaluate a clinical relevance the difference in infection rates will be analysed and interpreted numerically.

CONTACTS AND LOCATIONS:
Overall Officials: William JS Aston, MBBSMRCSFRCS, Principal Investigator — Royal National Orthopaedic Hospital
Locations (1):
- Royal National Orthopaedic Hospital, Stanmore, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be made available as all patient data is anonymised and therefore can not be traced back to individual patients

REFERENCES:
- [Background] Wafa H, Grimer RJ, Reddy K, Jeys L, Abudu A, Carter SR, Tillman RM. Retrospective evaluation of the incidence of early periprosthetic infection with silver-treated endoprostheses in high-risk patients: case-control study. Bone Joint J. 2015 Feb;97-B(2):252-7. doi: 10.1302/0301-620X.97B2.34554. PMID 25628291